CLINICAL TRIAL: NCT02685358
Title: An RCT of a Primary Care-Based PTSD Intervention: Clinician-Supported PTSD Coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 14-288; HX-001790-1 (Other Grant/Funding Number: U.S. Department of Veterans Affairs, HSR&D)
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress Disorders, Post-traumatic; Primary Health Care; Mobile Applications; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Clinician-Supported PTSD Coach (CS PTSD Coach) consists of four 20-30 minute sessions focused on instructions for using the PTSD Coach app, setting symptom reductions goals, and assigning specific PTSD Coach activities (i.e., assessments, management strategies, psycho-educational readings) for completion between sessions. PC-MHI providers deliver CS PTSD Coach using a treatment manual, which was developed and piloted by the PIs. Session 1 will be face-to-face and sessions 2-4 may be face-to-face or by phone, depending on patient preference. To help participants overcome treatment barriers psycho-education about treatment options are provided and active problems solving is encouraged. Specific next steps for treatment or self-management are developed collaboratively, typically in session 4. After session 4, Participants are encouraged to continue using PTSD Coach and have access to the research version of the app until the 24-week follow-up.
Who Masked: Outcomes Assessor
Masking Description: The CAPS-5 will be administered via phone by a central assessor, blind to condition, at baseline and post-treatment and will be the primary measure of change in PTSD symptom severity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinician-Supported PTSD Coach (Experimental): Clinician-supported PTSD Coach is primary care-based treatment. In this treatment a primary care mental health clinician guides patients in using the PTSD Coach mobile app to learn about PTSD symptoms, treatment options, and strategies to cope with common PTSD-related concerns. It consisted of 4 brief sessions over 8 weeks.
  Interventions: Behavioral: Clinician-Supported PTSD Coach
- Primary Care Mental Health Integrated Care as Usual (Active Comparator): Existing primary care mental health integrated treatment will serve as the comparison condition
  Interventions: Behavioral: Primary Care Mental Health Integrated Care as Usual

INTERVENTIONS:
Behavioral: Clinician-Supported PTSD Coach — Clinician-supported PTSD Coach is primary care-based treatment. In this treatment a primary care mental health clinician guides patients in using the PTSD Coach mobile app to learn about PTSD symptoms, treatment options, and strategies to cope with common PTSD-related concerns. It consists of 4 brief sessions over 8 weeks.
  Arms: Clinician-Supported PTSD Coach
Behavioral: Primary Care Mental Health Integrated Care as Usual — Existing primary care mental health integrated treatment will serve as the comparison condition
  Arms: Primary Care Mental Health Integrated Care as Usual

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is an often severe and frequently disabling condition. It is associated with compromised health, early mortality, and substantial economic costs. PTSD is common in VA primary care patients; however, brief, effective treatments for PTSD are not available in the primary care setting. Instead, patients with PTSD are referred to mental health settings, yet many patients do not accept these referrals or do not adequately engage in such services. Thus, this project seeks to improve health care for Veterans by testing the effectiveness of a primary care-based treatment called clinician-supported PTSD Coach. In this treatment a primary care mental health clinician guides patients in using the PTSD Coach mobile app to learn about PTSD symptoms, treatment options, and strategies to cope with common PTSD-related concerns. If this treatment is found to be effective at reducing PTSD symptoms and increasing use of mental health care, it will provide a tremendous benefit to Veterans with PTSD seen in VA primary care.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is an often severe and frequently disabling condition. It is associated with compromised health, early mortality, and substantial economic costs. PTSD is common in VA primary care patients; however, brief, effective treatments for PTSD are not available in the primary care setting. Instead, patients with PTSD are referred to mental health settings, yet many patients do not accept these referrals or do not adequately engage in such services. Thus, this project represents a unique opportunity to improve health care for Veterans by examining the effectiveness of a primary care-based treatment called Clinician-Supported PTSD Coach. In this treatment a primary care mental health clinician guides patients in using the PTSD Coach mobile app to learn about PTSD symptoms, treatment options, and strategies to cope with common PTSD-related concerns. This randomized clinical trial will enroll and treat 260 VA primary care patients (female and male) who have PTSD and are not currently being treated for it. Commonly used, well-established clinical interviews and self-report measures will be used to assess important clinical outcomes. If this direct treatment is found to be effective at reducing PTSD symptoms and increasing use of mental health care, it will provide a tremendous benefit to Veterans with PTSD seen in VA primary care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in primary care within the VA Syracuse and Palo Alto healthcare systems reporting 33 on the PTSD Checklist-5 (PCL-5) and a traumatic event on the Criterion A screener

Exclusion Criteria:

* Patients will be excluded if they demonstrate symptoms that would not allow them to actively engage in the CS PTSD Coach, i.e.,

  * gross cognitive impairment
* Current symptoms of mania or psychosis or who have more pressing concerns that need to be addressed first, i.e.,

  * suicide attempt in the last two months or current intent to commit suicide
* Patients with recent suicide attempts or intent are eligible to be enrolled follow the receipt of suicide prevention services
* The investigators will also exclude patients that are already receiving psychotherapy or MH counseling for PTSD outside of PC
* Started or changed the dose of a psychotropic medication for PTSD in the last two months that was prescribed outside of VA PC
* Voice a preference to be directly referred to MH specialty care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Kuhn, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Possemato K, Johnson E, Barrie K, Ghaus S, Noronha D, Wade M, Greenbaum MA, Rosen C, Cloitre M, Owen J, Jain S, Beehler G, Prins A, Seal K, Kuhn E. A Randomized Clinical Trial of Clinician-Supported PTSD Coach in VA Primary Care Patients. J Gen Intern Med. 2023 Jul;38(Suppl 3):905-912. doi: 10.1007/s11606-023-08130-6. Epub 2023 Mar 17. PMID 36932268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Started | 115 | 119
Completed | 100 | 112
Not Completed | 15 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual | Total
Number analyzed (Participants) | 115 | 119 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.04 (15.40) | 51.75 (15.47) | 50.92 (15.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 101 | 110 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 105 | 105 | 210
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 86 | 81 | 167
  Race: African American | 14 | 20 | 34
  Race: Asian/Pacific American | 6 | 6 | 12
  Race: Native American | 2 | 3 | 5
  Race: Multiracial | 4 | 7 | 11
  Race: Unknown or Missing | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 115 | 119 | 234
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — The CAPS-5 is a 30-item clinical interview that assesses the 20 DSM-5 PTSD symptoms. Scores on the CAPS-5 can range from 0 to 80, with higher scores reflecting worse PTSD symptom severity. In this study, clinician-rated PTSD symptom severity were based on blind assessor ratings.
  units on a scale | 28.52 (10.40) | 30.01 (10.36) | 29.28 (10.38)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The CAPS-5 is a 30-item clinical interview that assesses the 20 DSM-5 PTSD symptoms. Scores on the CAPS-5 can range from 0 to 80, with higher scores reflecting worse PTSD symptom severity. In this study, clinician-rated PTSD symptom severity were based on blind assessor ratings.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale | 28.52 (0.97) | 30.01 (0.95)

2. Primary Outcome: Hospital Administrative Data Showing 2 Mental Health Visits Completed
Description: Hospital administrative data will be examined to determine if the participant completed 2 visits to any specialty mental health clinic during the follow-up period.
Time Frame: 16 and 24 weeks
Population: For this outcome, only participants continuing to report significant PTSD symptoms (i.e., at or above the PCL-5 clinical cut score of 33) at 8 weeks were included. Per the protocol, these participants were offered a referral to specialty mental health treatment for PTSD.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 59 | 83
Participants | 21 | 20

3. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure assessing how much respondents have been bothered by DSM-5 PTSD symptoms in the past month. Scores can range from 0 to 80 with higher scores reflecting worse PTSD symptom severity.
Time Frame: Baseline, 8 week, 16 week, 24 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale
  Baseline | 46.30 (1.05) | 47.18 (1.03)
  8-week | 36.34 (1.2) | 40.68 (1.15)
  16-week | 35.42 (1.43) | 38.99 (1.35)
  24-week | 34.61 (1.69) | 38.05 (1.58)

4. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is a widely used 8-item self-report measure assessing patient satisfaction with care. Scores can range from 8 to 32 with higher scores reflecting greater satisfaction.
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale | 27.10 (3.73) | 24.60 (4.82)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: A 9-item self-report instrument used to assess depression severity. Items are scored 0 to 3, with the total score being the sum of the 9 items which can range from 0 as the minimum value to 27 as the maximum value. Higher scores indicate greater depression severity, with a score of 10 or greater indicating probable major depression, and scores of 20 or more severe major depression.
Time Frame: Baseline, 8 week, 16 week, 24 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale
  Baseline | 12.51 (.48) | 13.63 (.47)
  8-week | 11.03 (.50) | 12.12 (.48)
  16-week | 10.79 (.55) | 11.80 (.52)
  24-week | 10.22 (.61) | 11.30 (.57)

6. Secondary Outcome: WHOQOL-BREF Psychological Health Subscale
Description: The psychological health (6 items) subscale of the WHOQOL-BREF was used to assess the broader effects of the intervention on quality of life. Scores on this subscales range from 0-30 with higher scores reflecting better quality of life.
Time Frame: Baseline, 8 week, 16 week, 24 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale
  Baseline Psych Subscale | 17.82 (.35) | 17.51 (.34)
  8-week Psych Subscale | 18.16 (.37) | 17.50 (.35)
  16-week Psych Subscale | 18.04 (.39) | 17.65 (.37)
  24-week Psych Subscale | 18.29 (.42) | 17.47 (.40)

7. Secondary Outcome: WHOQOL-BREF Social Relationships Subscale
Description: The social relationships (3 items) subscale of the WHOQOL-BREF was used to assess the broader effects of the intervention on quality of life. Scores on this subscales range from 0-15 with higher scores reflecting better quality of life.
Time Frame: Baseline, 8 week, 16 week, 24 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
Number analyzed (Participants) | 115 | 119
score on a scale
  Baseline Social Subscale | 8.88 (.24) | 8.56 (.23)
  8-week Social Subscale | 9.31 (.24) | 8.71 (.23)
  16-week Social Subscale | 9.23 (.26) | 8.58 (.24)
  24-week Social Subscale | 9.01 (.27) | 8.40 (.25)

ADVERSE EVENTS:
Time Frame: For each enrolled participant, adverse event data was collected for the duration of their study participation, which was 24 weeks.
Arm/Group | Clinician-Supported PTSD Coach | Primary Care Mental Health Integrated Care as Usual
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/115 | 1/119
Other Adverse Events (participants affected / at risk) | 1/115 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician-Supported PTSD Coach (N=115) | Primary Care Mental Health Integrated Care as Usual (N=119)
Emergency Department Visit (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — The participant presented to community ER and was discharged the next day with right leg deep vein thrombosis (DVT, blood clot). Scheduled to follow up with the Syracuse VA.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician-Supported PTSD Coach (N=115) | Primary Care Mental Health Integrated Care as Usual (N=119)
Acute anger (Psychiatric disorders) | 1 (1) | 0 (0) — Participant became angry during the Clinician Administered PTSD Interview. The interviewer ended the assessment early. The participant was thanked for his time completing the portions of the assessment he did participate in.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02685358/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT02685358/SAP_001.pdf